CLINICAL TRIAL: NCT01743755
Title: Santeon-CAP; Dexamethasone in Community-acquired Pneumonia.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Collaborators: Canisius-Wilhelmina Hospital (Other); Onze Lieve Vrouw Hospital (Other); Catharina Ziekenhuis Eindhoven (Other); Maasstad Hospital (Other)
Responsible Party: Principal Investigator, Dr. WJW Bos, Principal Investigator, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Santeon-CAP; 2011-004566-14 (EudraCT Number)
Record Dates: First submitted 2012-11-22; First posted 2012-12-06 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Community-acquired Pneumonia
Keywords: Community-acquired pneumonia; Dexamethasone; Corticosteroid
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Active Comparator)
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Placebo tablet, once daily for four consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone tablet 6 mg, once daily for four consecutive days
  Arms: Dexamethasone
Drug: Placebo — Placebo tablet, once daily for four consecutive days
  Arms: Placebo

SUMMARY:
The present study is designed to investigate the beneficial effects of adjunctive dexamethasone therapy in patients admitted with community-acquired pneumonia, additionally aiming at assessing what patients benefit from dexamethasone treatment mostly. A large multicenter study will be conducted comparing a 4 days dexamethasone 6 mg per os course with placebo in 600 patients and with predefined subgroup analyses planned.

DETAILED DESCRIPTION:
Community-acquired pneumonia (CAP) is a common infection. Approximately 20 percent of all episodes of pneumonia result in hospitalization. It is the leading cause of community-acquired infection requiring intensive care unit (ICU) admission. In pulmonary infections, the release of cytokines and other inflammatory mediators from alveolar macrophages serves as a mechanism by which invading pathogens are eliminated. However, this reaction of the innate immune system can be potentially harmful when excessive release of circulating inflammatory cytokines causes damage to the patient, particularly the lung. Interest in the role of corticosteroids in the pathophysiology of critical illness has existed since the early part of the 20th century. On ICU, early treatment with corticosteroids to attenuate systemic inflammation is widespread. At the same time, outside the ICU little evidence is available on the effect of treatment with corticosteroids in patients diagnosed with CAP. Theoretically, early initiated administration of corticosteroids in the course of a CAP can lower systemic and pulmonary inflammation. This may lead to earlier resolution of pneumonia and a reduction of complications (sepsis, mortality).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Chest radiograph showing new opacities.

In combination with two of the following findings:

* Cough
* Production of sputum
* Temp >38,0 °C or <36,0 °C
* Audible abnormalities by chest examination compatible with pneumonia
* Leukocytosis (>10.000 cells/mm3), leftward shift (>10%) or leucopenia (<4000 cells/mm3)
* C-reactive protein > 15 mg/l (three fold higher than the upper limit of normal)

Exclusion Criteria:

* Immunocompromised patients:
* Patients with a known congenital or acquired immunodeficiency.
* Patients who received chemotherapy less than 6 weeks ago.
* Patients who received corticosteroids in the last 6 weeks.
* Patients who received immunosuppressive medication in the last 6 weeks (e.g. cyclosporin, cyclophosphamide, azathioprine).
* Patients with chronic obstructive pulmonary disease who are on systemic corticosteroids.
* Patients who require intensive care unit treatment.
* Patients with tropical worm infection.
* Patients with dexamethasone intolerance.
* Pregnant and breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2012-12; Primary Completion 2018-07-13 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Hospital admission (= day 1 = timepoint at which patient presents in hospital) until hospital discharge; participants will be followed for the duration of hospital stay, an expected average of 1 week.
  Discharge date will be the date on which the patient is clinically ready to be discharged (which means days of hospital stay on basis of social indication will be excluded from analyses). Median length of stay in an earlier CAP study performed in the St. Antonius Hospital in Nieuwegein was 6.5 days, thus patients will be followed during an expected average of 1 week.

SECONDARY OUTCOMES:
Mortality | day 30
  30 days after hospital admission (=day 1) the patient will visit the hospital for a out-patient visit. At that time, patient's status will be recorded.
ICU admission | hospital admission (=day 1) until hospital discharge; participants will be followed for the duration of hospital stay, an expected average of 1 week.
  In the period the patient is admitted to the hospital, admission to the intensive care unit will be recorded (yes/no and specific date).

OTHER OUTCOMES:
Mortality | Day 365
  One year after admission patient's status will be recorded.
S. pneumoniae prevalence | Hospital admission (= day 1)
  To study the prevalence of different S. pneumoniae serotypes in The Netherlands (based on the serotype distribution of isolated strains as well as the increase of serotype specific antibodies). Serotyping will be performed in a bloodsample taken on the day of admission.
Renal damage | Admission (=day 1) and day 30 (outpatient visist)
  To study acute renal damage, and its effect on outcome, in patients with CAP. A urine sample will be taken on the day of admission, on day 4 and on the outpatient visit at day 30.
Cost-effectiveness | Hospital discharge; participants will be followed for the duration of hospital stay, an expected average of 1 week.
  To study the cost-effectiveness of dexamethasone and outcome of CAP. Resource utilization will be acquired for the entire period of hospital stay for each individual patient.
Post-infectious fatigue | Day 30 and day 90
  To study post-infectious fatigue that occurs in certain patients after a CAP episode. On day 1, day 4, day of discharge, and 30 and 90 days after admission, the patient will be asked to fill in the EQ-5D questionnaire. Furthermore, on day 4, 30 and 90 days after admission, the patient will be asked to fill in the RAND-36 questionnaire.
Pathogenesis of CAP at respiratory mucosa | Day of admission (=day 1) and day 30 (outpatient visit)
  To study the pathogenesis of CAP at the respiratory mucosa (this will be done in two of the four study centra). At the day of hospital admission a nasopharyngeal swab will be taken to determine aetiology of the respiratory mucose. 30 days after admission (during the outpatient visit) another nasopharyngeal swab will be taken to explore changes.
Predefined subgroup analysis of length of stay | Hospital discharge; participants will be followed for the duration of hospital stay, an expected average of 1 week.
  To study what patients admitted with CAP benefit most from dexamethasone therapy, based on predefined subgroup analysis with:
  * disease severity score (PSI 1-3 vs. PSI 4-5);
  * C-reactive protein level at admission;
  * causative microorganism (Pneumococcus urinary antigen test positive vs. negative);
  * cytokine response (IL-6 and IL-10) over time;
  * cortisol level over time;
  * procalcitonin over time;
  * vitamin D level on admission.

CONTACTS AND LOCATIONS:
Overall Officials: Willem Jan Bos, MD, PhD, Principal Investigator — St. Antonius Hospital; Jan Grutters, Prof, MD, Principal Investigator — St. Antonius Hospital; Rob Janssen, MD, PhD, Principal Investigator — Canisius-Wilhelmina Hospital; Frank Smeenk, MD, PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven; Paul Bresser, MD, PhD, Principal Investigator — Onze Lieve Vrouwen Gasthuis; Stijn Konings, MD, PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven; Willem Blok, MD, PhD, Principal Investigator — Onze Lieve Vrouwen Gasthuis
Locations (4):
- Netherlands (4):
  - Canisius Wilhelmina Hospital, Nijmegen, Gelderland
  - Catharina hospital Eindhoven, Eindhoven, North Brabant
  - OLVG, Amsterdam, North Holland
  - St. Antonius Hospital, Nieuwegein, Utrecht

REFERENCES:
- [Background] Meijvis SC, Hardeman H, Remmelts HH, Heijligenberg R, Rijkers GT, van Velzen-Blad H, Voorn GP, van de Garde EM, Endeman H, Grutters JC, Bos WJ, Biesma DH. Dexamethasone and length of hospital stay in patients with community-acquired pneumonia: a randomised, double-blind, placebo-controlled trial. Lancet. 2011 Jun 11;377(9782):2023-30. doi: 10.1016/S0140-6736(11)60607-7. Epub 2011 Jun 1. PMID 21636122
- [Derived] Wittermans E, Vestjens SMT, Spoorenberg SMC, Blok WL, Grutters JC, Janssen R, Rijkers GT, Smeenk FWJM, Voorn GP, van de Garde EMW, Bos WJW; Santeon-CAP Study Group; Members of the Santeon-CAP Study Group. Adjunctive treatment with oral dexamethasone in non-ICU patients hospitalised with community-acquired pneumonia: a randomised clinical trial. Eur Respir J. 2021 Aug 12;58(2):2002535. doi: 10.1183/13993003.02535-2020. Print 2021 Aug. PMID 33446608
- [Derived] Vestjens SMT, Wittermans E, Spoorenberg SMC, Grutters JC, van Ruitenbeek CA, Voorn GP, Bos WJW, van de Garde EMW. Inter-hospital variation in the utilization of diagnostics and their proportionality in the management of adult community-acquired pneumonia. Pneumonia (Nathan). 2018 Dec 25;10:15. doi: 10.1186/s41479-018-0059-0. eCollection 2018. PMID 30603378